CLINICAL TRIAL: NCT05081284
Title: Clinical Outcomes of Immediate Implants With or Without a Volume-stable Collagen Matrix: a Randomized Controlled Clinical Trial
Brief Title: Clinical Outcomes of Immediate Implants With or Without a Volume-stable Collagen Matrix
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonio Barone, Professor, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19228
Record Dates: First submitted 2021-09-20; First posted 2021-10-18 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Edentulous Alveolar Ridge
Keywords: Soft tissue augmentation; Immediate implant; Collagen matrix

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Immediate implant insertion in fresh-extraction site, will be performed. Peri-implant bone defect will be grafted with a deproteinized bovine bone mineral with 10% collagen and covered with a collagen matrix. After the surgical procedures, each implant will receive a healing abutment until prosthetic restorative procedures.
- Test Group (Experimental): Immediate implant insertion in fresh-extraction site, will be performed. Peri-implant bone defect will be grafted with a deproteinized bovine bone mineral with 10% collagen and covered with a collagen matrix, and then a volume-stable collagen matrix will be buccally inserted with a split-thickness flap preparation. Subsequently, the collagen matrix graft will be stabilized with a horizontal mattress suture to the buccal flap. After the surgical procedures, each implant will receive healing abutment connection until the prosthetic restorative procedures
  Interventions: Device: Volume-stable collagen matrix Geistlich Fibro-Gide®

INTERVENTIONS:
Device: Volume-stable collagen matrix Geistlich Fibro-Gide® — After tooth extraction and implant insertion the Test group will receive a soft tissue augmentation on the buccal side oh the implant. an envelop flap will be raised and a volume-stable collagen graft will be stabilized with sutures.
  Control group will not receive soft tissue augmentation.
  Other Names: Geistlich Fibro-Gide, G1 039446 0086 Rev. 00 G7 16 07 39446 073
  Arms: Test Group

SUMMARY:
The purpose of this study is to evaluate the soft tissue clinical results in patients that received, or not, a soft tissue augmentation around dental implant inserted immediately after the extraction.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a screening period to determinate eligibility for study entry. Patients who meet eligibility requirements will be randomized in this single blinded(investigator) study.

Group (Test) will receive immediate implant after extraction and a soft tissue augmentation with a collagen matrix.

Group (Control) will receive only immediate implant after extraction without soft tissue augmentation.

ELIGIBILITY:
Inclusion Criteria:

- Presence of a single failing tooth in the esthetic region (second premolar to contralateral second premolar), the adjacent teeth should be present and without any dental pathologies.

Exclusion Criteria:

* Patients who are heavy smokers (more than 10 cigarettes/day);
* Patients who suffer from any systemic diseases that could negatively influence wound healing;
* Patients who received head and neck radiation treatment;
* Patients who have a full contraindication to implant surgery;
* Patients who have uncontrolled periodontal disease;
* Patients who show a full mouth plaque and bleeding score higher than 25%;
* Patients who have deficient extraction sockets according to the classification of Juodzbalys et al. 2008.
* Patients with known allergy, sensitivity or intolerance to collagen
* Patients who are pregnant or who are breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Soft Tissue Thickness (STT) | T0a: baseline before surgery
  Measured at 3 and 6 mm from the free gingival margin using a 15-endodontic file and a rubber disk. The file will advance perpendicularly through the soft tissue until the first point of bone contact. Thickness will be measured to the nearest 0.1 mm using a caliper. The rubber disk stop will be then placed in tight contact with the soft tissue surface and fixed with a drop of cyanocrylic adhesive. After file removal, the distance between file tip and the silicon stop will be measured using a digital caliper with 0.01 mm of accuracy. (Cairo et al. 2017; Bittner et al. 2020)
Soft Tissue Thickness (STT) | T0b: baseline after surgery
  Measured at 3 and 6 mm from the free gingival margin using a 15-endodontic file and a rubber disk. The file will advance perpendicularly through the soft tissue until the first point of bone contact. Thickness will be measured to the nearest 0.1 mm using a caliper. The rubber disk stop will be then placed in tight contact with the soft tissue surface and fixed with a drop of cyanocrylic adhesive. After file removal, the distance between file tip and the silicon stop will be measured using a digital caliper with 0.01 mm of accuracy. (Cairo et al. 2017; Bittner et al. 2020)
Soft Tissue Thickness (STT) | T2: 12 months after implant placement
  Measured at 3 and 6 mm from the free gingival margin using a 15-endodontic file and a rubber disk. The file will advance perpendicularly through the soft tissue until the first point of bone contact. Thickness will be measured to the nearest 0.1 mm using a caliper. The rubber disk stop will be then placed in tight contact with the soft tissue surface and fixed with a drop of cyanocrylic adhesive. After file removal, the distance between file tip and the silicon stop will be measured using a digital caliper with 0.01 mm of accuracy. (Cairo et al. 2017; Bittner et al. 2020)

SECONDARY OUTCOMES:
Vertical position of soft tissue (VPS) | T0a: baseline before surgery
  A tooth-supported Essix stent will be used to record the distance from three reference marks (mesial papilla, midbuccal margin, and distal papilla) to the free gingival margin using a color-coded probe (15mm, UNC). The same stent will be used for measurements at the different follow-up visits. (Bittner et al. 2020)
Vertical position of soft tissue (VPS) | T0b: baseline after surgery
  A tooth-supported Essix stent will be used to record the distance from three reference marks (mesial papilla, midbuccal margin, and distal papilla) to the free gingival margin using a color-coded probe (15mm, UNC). The same stent will be used for measurements at the different follow-up visits. (Bittner et al. 2020)
Vertical position of soft tissue (VPS) | T1: 2 weeks after crown delivery, 4 months from surgery
  A tooth-supported Essix stent will be used to record the distance from three reference marks (mesial papilla, midbuccal margin, and distal papilla) to the free gingival margin using a color-coded probe (15mm, UNC). The same stent will be used for measurements at the different follow-up visits. (Bittner et al. 2020)
Vertical position of soft tissue (VPS) | T2: 12 months after surgery
  A tooth-supported Essix stent will be used to record the distance from three reference marks (mesial papilla, midbuccal margin, and distal papilla) to the free gingival margin using a color-coded probe (15mm, UNC). The same stent will be used for measurements at the different follow-up visits. (Bittner et al. 2020)
Vertical position of soft tissue (VPS) | T3: 24 months after surgery
  A tooth-supported Essix stent will be used to record the distance from three reference marks (mesial papilla, midbuccal margin, and distal papilla) to the free gingival margin using a color-coded probe (15mm, UNC). The same stent will be used for measurements at the different follow-up visits. (Bittner et al. 2020)
Vertical position of soft tissue (VPS) | T4: 36 months after surgery
  A tooth-supported Essix stent will be used to record the distance from three reference marks (mesial papilla, midbuccal margin, and distal papilla) to the free gingival margin using a color-coded probe (15mm, UNC). The same stent will be used for measurements at the different follow-up visits. (Bittner et al. 2020)
Assessment of the linear volumetric changes | T0a: baseline before surgery
  Impressions of the grafted sites will be taken including at least the two neighboring teeth and using a silicone impression material. Dental stone casts will be fabricated and optically scanned with a desktop 3D scanner. Digital models of each time-point per patient will be captured as stereolithography (STL) files. The images of the baseline and follow-up datasets will be superimposed and matched using the best-fit algorithm at the adjacent tooth surfaces. After definition of specific regions of interest (ROI), the software will calculated the volumetric changes measured in mm, which will correspond to the mean distance between the three surfaces representing the evaluated time-points. One buccal ROI will be defined: a trapezoid shape area between the gingival margins of the adjacent teeth, the mucogingival junction as apical and the interproximal areas as lateral borders. The measured will be kept constant in each patient and site over time. (Zeltner 2017)
Assessment of the linear volumetric changes | T1: 2 weeks after crown delivery, 4 months from surgery
  Impressions of the grafted sites will be taken including at least the two neighboring teeth and using a silicone impression material. Dental stone casts will be fabricated and optically scanned with a desktop 3D scanner. Digital models of each time-point per patient will be captured as stereolithography (STL) files. The images of the baseline and follow-up datasets will be superimposed and matched using the best-fit algorithm at the adjacent tooth surfaces. After definition of specific regions of interest (ROI), the software will calculated the volumetric changes measured in mm, which will correspond to the mean distance between the three surfaces representing the evaluated time-points. One buccal ROI will be defined: a trapezoid shape area between the gingival margins of the adjacent teeth, the mucogingival junction as apical and the interproximal areas as lateral borders. The measured will be kept constant in each patient and site over time. (Zeltner 2017)
Assessment of the linear volumetric changes | T2: 12 months after surgery
  Impressions of the grafted sites will be taken including at least the two neighboring teeth and using a silicone impression material. Dental stone casts will be fabricated and optically scanned with a desktop 3D scanner. Digital models of each time-point per patient will be captured as stereolithography (STL) files. The images of the baseline and follow-up datasets will be superimposed and matched using the best-fit algorithm at the adjacent tooth surfaces. After definition of specific regions of interest (ROI), the software will calculated the volumetric changes measured in mm, which will correspond to the mean distance between the three surfaces representing the evaluated time-points. One buccal ROI will be defined: a trapezoid shape area between the gingival margins of the adjacent teeth, the mucogingival junction as apical and the interproximal areas as lateral borders. The measured will be kept constant in each patient and site over time. (Zeltner 2017)
Assessment of the linear volumetric changes | T3: 24 months after surgery
  Impressions of the grafted sites will be taken including at least the two neighboring teeth and using a silicone impression material. Dental stone casts will be fabricated and optically scanned with a desktop 3D scanner. Digital models of each time-point per patient will be captured as stereolithography (STL) files. The images of the baseline and follow-up datasets will be superimposed and matched using the best-fit algorithm at the adjacent tooth surfaces. After definition of specific regions of interest (ROI), the software will calculated the volumetric changes measured in mm, which will correspond to the mean distance between the three surfaces representing the evaluated time-points. One buccal ROI will be defined: a trapezoid shape area between the gingival margins of the adjacent teeth, the mucogingival junction as apical and the interproximal areas as lateral borders. The measured will be kept constant in each patient and site over time. (Zeltner 2017)
Assessment of the linear volumetric changes | T4: 36 months after surgery
  Impressions of the grafted sites will be taken including at least the two neighboring teeth and using a silicone impression material. Dental stone casts will be fabricated and optically scanned with a desktop 3D scanner. Digital models of each time-point per patient will be captured as stereolithography (STL) files. The images of the baseline and follow-up datasets will be superimposed and matched using the best-fit algorithm at the adjacent tooth surfaces. After definition of specific regions of interest (ROI), the software will calculated the volumetric changes measured in mm, which will correspond to the mean distance between the three surfaces representing the evaluated time-points. One buccal ROI will be defined: a trapezoid shape area between the gingival margins of the adjacent teeth, the mucogingival junction as apical and the interproximal areas as lateral borders. The measured will be kept constant in each patient and site over time. (Zeltner 2017)
Pink Esthetic Score (PES) | T1: 2 weeks after crown delivery, 4 months from surgery
  PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft- tissue contour, alveolar process deficiency, soft-tissue colour and texture. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score. The papillae values will be evaluated for completeness, incompleteness or absence. Other variables will be assessed by comparison with a reference tooth. The highest possible score reflecting a perfect match of the peri-implant soft tissue with that of the reference tooth will be 14. (Furhauser et al. 2005)
Pink Esthetic Score (PES) | T2: 12 months after surgery
  PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft- tissue contour, alveolar process deficiency, soft-tissue colour and texture. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score. The papillae values will be evaluated for completeness, incompleteness or absence. Other variables will be assessed by comparison with a reference tooth. The highest possible score reflecting a perfect match of the peri-implant soft tissue with that of the reference tooth will be 14. (Furhauser et al. 2005)
Pink Esthetic Score (PES) | T3: 24 months after surgery
  PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft- tissue contour, alveolar process deficiency, soft-tissue colour and texture. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score. The papillae values will be evaluated for completeness, incompleteness or absence. Other variables will be assessed by comparison with a reference tooth. The highest possible score reflecting a perfect match of the peri-implant soft tissue with that of the reference tooth will be 14. (Furhauser et al. 2005)
Pink Esthetic Score (PES) | T4: 36 months after surgery
  PES is based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft- tissue contour, alveolar process deficiency, soft-tissue colour and texture. Each variable will be assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score. The papillae values will be evaluated for completeness, incompleteness or absence. Other variables will be assessed by comparison with a reference tooth. The highest possible score reflecting a perfect match of the peri-implant soft tissue with that of the reference tooth will be 14. (Furhauser et al. 2005)
Papillae index (PI) | T0a: baseline before surgery
  The statuses of the mesial and distal papilla will be assessed using the Papillae index (from 0 to 3). (Jemt et al. 1997)
Papillae index (PI) | T0b: baseline after surgery
  The statuses of the mesial and distal papilla will be assessed using the Papillae index (from 0 to 3). (Jemt et al. 1997)
Papillae index (PI) | T1: 2 weeks after crown delivery, 4 months from surgery
  The statuses of the mesial and distal papilla will be assessed using the Papillae index (from 0 to 3). (Jemt et al. 1997)
Papillae index (PI) | T2: 12 months after surgery
  The statuses of the mesial and distal papilla will be assessed using the Papillae index (from 0 to 3). (Jemt et al. 1997)
Papillae index (PI) | T3: 24 months after surgery
  The statuses of the mesial and distal papilla will be assessed using the Papillae index (from 0 to 3). (Jemt et al. 1997)
Papillae index (PI) | T4: 36 months after surgery
  The statuses of the mesial and distal papilla will be assessed using the Papillae index (from 0 to 3). (Jemt et al. 1997)
Width of keratinized tissue (WKT) | T0a: baseline before surgery
  WKT will be measured, with a periodontal probe (mm), mid-facially from the gingival margin to the muco-gingival junction of the intended extracted tooth or the implant supported restoration.
Width of keratinized tissue (WKT) | T1: 2 weeks after crown delivery, 4 months from surgery
  WKT will be measured, with a periodontal probe (mm), mid-facially from the gingival margin to the muco-gingival junction of the intended extracted tooth or the implant supported restoration.
Width of keratinized tissue (WKT) | T2: 12 months after surgery
  WKT will be measured, with a periodontal probe (mm), mid-facially from the gingival margin to the muco-gingival junction of the intended extracted tooth or the implant supported restoration.
Width of keratinized tissue (WKT) | T3: 24 months after surgery
  WKT will be measured, with a periodontal probe (mm), mid-facially from the gingival margin to the muco-gingival junction of the intended extracted tooth or the implant supported restoration.
Width of keratinized tissue (WKT) | T4: 36 months after surgery
  WKT will be measured, with a periodontal probe (mm), mid-facially from the gingival margin to the muco-gingival junction of the intended extracted tooth or the implant supported restoration.
Peri-implant marginal bone level (MBL) | T0b: baseline after surgery
  MBL will be measured on intraoral radiographs at the mesial and distal aspects (m and d). It will be set as the distance between the reference point and the most apical point of contact between the implant surface and the bone. The reference point will be the fixture-abutment interface. Digital intraoral periapical radiographs will be taken using a parallel cone technique with digital sensor. A paralleling device and individualized bite blocks made of polyvinyl siloxane impression material will be used for the standardization of the X-ray geometry. Calibration will be performed using the known thread-pitch distance of the implants. Measurements will be taken to the nearest millimeter using computer software.
Peri-implant marginal bone level (MBL) | T1: 2 weeks after crown delivery, 4 months from surgery
  MBL will be measured on intraoral radiographs at the mesial and distal aspects (m and d). It will be set as the distance between the reference point and the most apical point of contact between the implant surface and the bone. The reference point will be the fixture-abutment interface. Digital intraoral periapical radiographs will be taken using a parallel cone technique with digital sensor. A paralleling device and individualized bite blocks made of polyvinyl siloxane impression material will be used for the standardization of the X-ray geometry. Calibration will be performed using the known thread-pitch distance of the implants. Measurements will be taken to the nearest millimeter using computer software.
Peri-implant marginal bone level (MBL) | T2: 12 months after surgery
  MBL will be measured on intraoral radiographs at the mesial and distal aspects (m and d). It will be set as the distance between the reference point and the most apical point of contact between the implant surface and the bone. The reference point will be the fixture-abutment interface. Digital intraoral periapical radiographs will be taken using a parallel cone technique with digital sensor. A paralleling device and individualized bite blocks made of polyvinyl siloxane impression material will be used for the standardization of the X-ray geometry. Calibration will be performed using the known thread-pitch distance of the implants. Measurements will be taken to the nearest millimeter using computer software.
Peri-implant marginal bone level (MBL) | T3: 24 months after surgery
  MBL will be measured on intraoral radiographs at the mesial and distal aspects (m and d). It will be set as the distance between the reference point and the most apical point of contact between the implant surface and the bone. The reference point will be the fixture-abutment interface. Digital intraoral periapical radiographs will be taken using a parallel cone technique with digital sensor. A paralleling device and individualized bite blocks made of polyvinyl siloxane impression material will be used for the standardization of the X-ray geometry. Calibration will be performed using the known thread-pitch distance of the implants. Measurements will be taken to the nearest millimeter using computer software.
Peri-implant marginal bone level (MBL) | T4: 36 months after surgery
  MBL will be measured on intraoral radiographs at the mesial and distal aspects (m and d). It will be set as the distance between the reference point and the most apical point of contact between the implant surface and the bone. The reference point will be the fixture-abutment interface. Digital intraoral periapical radiographs will be taken using a parallel cone technique with digital sensor. A paralleling device and individualized bite blocks made of polyvinyl siloxane impression material will be used for the standardization of the X-ray geometry. Calibration will be performed using the known thread-pitch distance of the implants. Measurements will be taken to the nearest millimeter using computer software.
Phenotype | T0a: baseline before surgery
  It will be based on the lack of transparency of a periodontal probe through the gingival margin when probing the buccal sulcus of the failing tooth (De Rouck et al. 2009).
Phenotype | T1: 2 weeks after crown delivery, 4 months from surgery
  It will be based on the lack of transparency of a periodontal probe through the gingival margin when probing the buccal sulcus of the failing tooth (De Rouck et al. 2009).
Phenotype | T2: 12 months after surgery
  It will be based on the lack of transparency of a periodontal probe through the gingival margin when probing the buccal sulcus of the failing tooth (De Rouck et al. 2009).
Phenotype | T3: 24 months after surgery
  It will be based on the lack of transparency of a periodontal probe through the gingival margin when probing the buccal sulcus of the failing tooth (De Rouck et al. 2009).
Phenotype | T4: 36 months after surgery
  It will be based on the lack of transparency of a periodontal probe through the gingival margin when probing the buccal sulcus of the failing tooth (De Rouck et al. 2009).
Probing pocket depth (PD) | T0a: baseline before surgery
  probing pocket depth using a manual periodontal probe at the mesio-buccal, mid-buccal, and disto-buccal and mid-palatal aspect. The distance measured from the base of the pocket to the most apical point on the gingival margin, expressed in millimeters (Mombelli et al., 1987).
Probing pocket depth (PD) | T1: 2 weeks after crown delivery, 4 months from surgery
  probing pocket depth using a manual periodontal probe at the mesio-buccal, mid-buccal, and disto-buccal and mid-palatal aspect.The distance measured from the base of the pocket to the most apical point on the gingival margin, expressed in millimeters (Mombelli et al., 1987).
Probing pocket depth (PD) | T2: 12 months after surgery
  probing pocket depth using a manual periodontal probe at the mesio-buccal, mid-buccal, and disto-buccal and mid-palatal aspect.The distance measured from the base of the pocket to the most apical point on the gingival margin, expressed in millimeters (Mombelli et al., 1987).
Probing pocket depth (PD) | T3: 24 months after surgery
  probing pocket depth using a manual periodontal probe at the mesio-buccal, mid-buccal, and disto-buccal and mid-palatal aspect.The distance measured from the base of the pocket to the most apical point on the gingival margin, expressed in millimeters (Mombelli et al., 1987).
Probing pocket depth (PD) | T4: 36 months after surgery
  probing pocket depth using a manual periodontal probe at the mesio-buccal, mid-buccal, and disto-buccal and mid-palatal aspect.The distance measured from the base of the pocket to the most apical point on the gingival margin, expressed in millimeters (Mombelli et al., 1987).
Modified Plaque Index (mPI) | T0a: baseline before surgery
  Modified Plaque Index (mPI) is a dental plaque scale as follows 0 = No plaque,
  1 = Separate flecks of plaque at the cervical margin;2 = Plaque can be seen by naked eye.3 = Abundance of soft matter. The lower the number the less plaque is present on the tooth. (Mombelli et al., 1987);
Modified Plaque Index (mPI) | T1: 2 weeks after crown delivery, 4 months from surgery
  Modified Plaque Index (mPI) is a dental plaque scale as follows 0 = No plaque,
  1 = Separate flecks of plaque at the cervical margin;2 = Plaque can be seen by naked eye.3 = Abundance of soft matter. The lower the number the less plaque is present on the tooth. (Mombelli et al., 1987);
Modified Plaque Index (mPI) | T2: 12 months after surgery
  Modified Plaque Index (mPI) is a dental plaque scale as follows 0 = No plaque,
  1 = Separate flecks of plaque at the cervical margin;2 = Plaque can be seen by naked eye.3 = Abundance of soft matter. The lower the number the less plaque is present on the tooth. (Mombelli et al., 1987);
Modified Plaque Index (mPI) | T3: 24 months after surgery
  Modified Plaque Index (mPI) is a dental plaque scale as follows 0 = No plaque,
  1 = Separate flecks of plaque at the cervical margin;2 = Plaque can be seen by naked eye.3 = Abundance of soft matter. The lower the number the less plaque is present on the tooth. (Mombelli et al., 1987);
Modified Plaque Index (mPI) | T4: 36 months after surgery
  Modified Plaque Index (mPI) is a dental plaque scale as follows 0 = No plaque,
  1 = Separate flecks of plaque at the cervical margin;2 = Plaque can be seen by naked eye.3 = Abundance of soft matter. The lower the number the less plaque is present on the tooth. (Mombelli et al., 1987);
Gingival bleeding on probing (BoP) | T0a: baseline before surgery
  Gingival bleeding on probing (BOP) using the modified sulcus bleeding index for implants. Scale equals 0 = No bleeding when periodontal probe is passed along the gingival margin;1 = Isolated bleeding spots visible;2 = Blood forms a confluent red line on the gingival margin;3 = Heavy or profuse bleeding. (Mombelli et al., 1987).
Gingival bleeding on probing (BoP) | T1: 2 weeks after crown delivery, 4 months from surgery
  Gingival bleeding on probing (BOP) using the modified sulcus bleeding index for implants. Scale equals 0 = No bleeding when periodontal probe is passed along the gingival margin;1 = Isolated bleeding spots visible;2 = Blood forms a confluent red line on the gingival margin;3 = Heavy or profuse bleeding. (Mombelli et al., 1987).
Gingival bleeding on probing (BoP) | T2: 12 months after surgery
  Gingival bleeding on probing (BOP) using the modified sulcus bleeding index for implants. Scale equals 0 = No bleeding when periodontal probe is passed along the gingival margin;1 = Isolated bleeding spots visible;2 = Blood forms a confluent red line on the gingival margin;3 = Heavy or profuse bleeding. (Mombelli et al., 1987).
Gingival bleeding on probing (BoP) | T3: 24 months after surgery
  Gingival bleeding on probing (BOP) using the modified sulcus bleeding index for implants. Scale equals 0 = No bleeding when periodontal probe is passed along the gingival margin;1 = Isolated bleeding spots visible;2 = Blood forms a confluent red line on the gingival margin;3 = Heavy or profuse bleeding. (Mombelli et al., 1987).
Gingival bleeding on probing (BoP) | T4: 36 months after surgery
  Gingival bleeding on probing (BOP) using the modified sulcus bleeding index for implants. Scale equals 0 = No bleeding when periodontal probe is passed along the gingival margin;1 = Isolated bleeding spots visible;2 = Blood forms a confluent red line on the gingival margin;3 = Heavy or profuse bleeding. (Mombelli et al., 1987).
Implant success | T1: 2 weeks after crown delivery, 4 months from surgery
  Implant failure and Implant success criteria will be recorded according to Buser et al.1990.
Implant success | T2: 12 months after surgery
  Implant failure and Implant success criteria will be recorded according to Buser et al.1990.
Implant success | T3: 24 months after surgery
  Implant failure and Implant success criteria will be recorded according to Buser et al.1990.
Implant success | T4: 36 months after surgery
  Implant failure and Implant success criteria will be recorded according to Buser et al.1990.
Biological and technical complication | T0a: baseline before surgery
  Complications from biological and technical nature (Pjetursson et al. 2012).
Biological and technical complication | T0b: baseline after surgery
  Complications from biological and technical nature (Pjetursson et al. 2012).
Biological and technical complication | T1: 2 weeks after crown delivery, 4 months from surgery
  Complications from biological and technical nature (Pjetursson et al. 2012).
Biological and technical complication | T2: 12 months after surgery
  Complications from biological and technical nature (Pjetursson et al. 2012).
Biological and technical complication | T3: 24 months after surgery
  Complications from biological and technical nature (Pjetursson et al. 2012).
Biological and technical complication | T4: 36 months after surgery
  Complications from biological and technical nature (Pjetursson et al. 2012).
Surgery time | T0a-b: baseline
  The surgery time will be recorded in both groups to the closest minute from the start of the first incision to the accomplishment of the last suture.
Patient satisfaction OHIP-14 | T0a: baseline before surgery
  The Oral Health Impact Profile (OHIP-14) is a questionnaire addressed the following domains: functional limitation, physical pain, psychological discomfort, physical disability, psycho- logical disability, social disability and handicap. These domains were evaluated by 2 questions each and scored by means of a 5-point Likert scale resulting in a total OHIP score ranging from 14 to 70 with higher scores being indicative of more discomfort in daily life. (Slade & Spencer, 1994)
Patient satisfaction OHIP-14 | T1: 2 weeks after crown delivery, 4 months from surgery
  The Oral Health Impact Profile (OHIP-14) is a questionnaire addressed the following domains: functional limitation, physical pain, psychological discomfort, physical disability, psycho- logical disability, social disability and handicap. These domains were evaluated by 2 questions each and scored by means of a 5-point Likert scale resulting in a total OHIP score ranging from 14 to 70 with higher scores being indicative of more discomfort in daily life. (Slade & Spencer, 1994)
Patient satisfaction OHIP-14 | T2: 12 months after surgery
  The Oral Health Impact Profile (OHIP-14) is a questionnaire addressed the following domains: functional limitation, physical pain, psychological discomfort, physical disability, psycho- logical disability, social disability and handicap. These domains were evaluated by 2 questions each and scored by means of a 5-point Likert scale resulting in a total OHIP score ranging from 14 to 70 with higher scores being indicative of more discomfort in daily life. (Slade & Spencer, 1994)
Patient satisfaction OHIP-14 | T3: 24 months after surgery
  The Oral Health Impact Profile (OHIP-14) is a questionnaire addressed the following domains: functional limitation, physical pain, psychological discomfort, physical disability, psycho- logical disability, social disability and handicap. These domains were evaluated by 2 questions each and scored by means of a 5-point Likert scale resulting in a total OHIP score ranging from 14 to 70 with higher scores being indicative of more discomfort in daily life. (Slade & Spencer, 1994)
Patient satisfaction OHIP-14 | T4: 36 months after surgery
  The Oral Health Impact Profile (OHIP-14) is a questionnaire addressed the following domains: functional limitation, physical pain, psychological discomfort, physical disability, psycho- logical disability, social disability and handicap. These domains were evaluated by 2 questions each and scored by means of a 5-point Likert scale resulting in a total OHIP score ranging from 14 to 70 with higher scores being indicative of more discomfort in daily life. (Slade & Spencer, 1994)
Patient satisfaction VAS | T0a: baseline before surgery
  Patients were asked to respond to the following question on a Visual analogic scale: "How satisfied are you with the overall aesthetic result?" and "How satisfied are you with the overall functional result?"."Most unsatisfied" and "most satisfied" were indicated as extremes on the 100-mm lines.
Patient satisfaction VAS | T1: 2 weeks after crown delivery, 4 months from surgery
  Patients were asked to respond to the following question on a Visual analogic scale: "How satisfied are you with the overall aesthetic result?" and "How satisfied are you with the overall functional result?"."Most unsatisfied" and "most satisfied" were indicated as extremes on the 100-mm lines.
Patient satisfaction VAS | T2: 12 months after surgery
  Patients were asked to respond to the following question on a Visual analogic scale: "How satisfied are you with the overall aesthetic result?" and "How satisfied are you with the overall functional result?"."Most unsatisfied" and "most satisfied" were indicated as extremes on the 100-mm lines.
Patient satisfaction VAS | T3: 24 months after surgery
  Patients were asked to respond to the following question on a Visual analogic scale: "How satisfied are you with the overall aesthetic result?" and "How satisfied are you with the overall functional result?"."Most unsatisfied" and "most satisfied" were indicated as extremes on the 100-mm lines.
Patient satisfaction VAS | T4: 36 months after surgery
  Patients were asked to respond to the following question on a Visual analogic scale: "How satisfied are you with the overall aesthetic result?" and "How satisfied are you with the overall functional result?"."Most unsatisfied" and "most satisfied" were indicated as extremes on the 100-mm lines.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Barone, DDS, Principal Investigator — University of Pisa
Locations (1):
- U.O. Odontostomatologia e Chirurgia del Cavo Orale, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cairo F, Barbato L, Tonelli P, Batalocco G, Pagavino G, Nieri M. Xenogeneic collagen matrix versus connective tissue graft for buccal soft tissue augmentation at implant site. A randomized, controlled clinical trial. J Clin Periodontol. 2017 Jul;44(7):769-776. doi: 10.1111/jcpe.12750. Epub 2017 Jun 29. PMID 28548210
- [Result] Bittner N, Planzos L, Volchonok A, Tarnow D, Schulze-Spate U. Evaluation of Horizontal and Vertical Buccal Ridge Dimensional Changes After Immediate Implant Placement and Immediate Temporization With and Without Bone Augmentation Procedures: Short-Term, 1-Year Results. A Randomized Controlled Clinical Trial. Int J Periodontics Restorative Dent. 2020 Jan/Feb;40(1):83-93. doi: 10.11607/prd.4152. PMID 31815977
- [Result] Zeltner M, Jung RE, Hammerle CH, Husler J, Thoma DS. Randomized controlled clinical study comparing a volume-stable collagen matrix to autogenous connective tissue grafts for soft tissue augmentation at implant sites: linear volumetric soft tissue changes up to 3 months. J Clin Periodontol. 2017 Apr;44(4):446-453. doi: 10.1111/jcpe.12697. Epub 2017 Feb 11. PMID 28107560
- [Result] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Result] Jemt T. Regeneration of gingival papillae after single-implant treatment. Int J Periodontics Restorative Dent. 1997 Aug;17(4):326-33. PMID 9497723
- [Result] De Rouck T, Eghbali R, Collys K, De Bruyn H, Cosyn J. The gingival biotype revisited: transparency of the periodontal probe through the gingival margin as a method to discriminate thin from thick gingiva. J Clin Periodontol. 2009 May;36(5):428-33. doi: 10.1111/j.1600-051X.2009.01398.x. PMID 19419444
- [Result] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Result] Buser D, Weber HP, Lang NP. Tissue integration of non-submerged implants. 1-year results of a prospective study with 100 ITI hollow-cylinder and hollow-screw implants. Clin Oral Implants Res. 1990 Dec;1(1):33-40. doi: 10.1034/j.1600-0501.1990.010105.x. PMID 2099210
- [Result] Pjetursson BE, Thoma D, Jung R, Zwahlen M, Zembic A. A systematic review of the survival and complication rates of implant-supported fixed dental prostheses (FDPs) after a mean observation period of at least 5 years. Clin Oral Implants Res. 2012 Oct;23 Suppl 6:22-38. doi: 10.1111/j.1600-0501.2012.02546.x. PMID 23062125
- [Result] van der Meulen MJ, Lobbezoo F, John MT, Naeije M. [Oral health impact profile. an instrument for measuring the impact of oral health on the quality of life]. Ned Tijdschr Tandheelkd. 2011 Mar;118(3):134-9. doi: 10.5177/ntvt.2011.03.10178. Dutch. PMID 21491763